CLINICAL TRIAL: NCT02222779
Title: Quantification of Transition Metals in Patients at the Cologne University Hospital
Brief Title: Quantification of Transition Metals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Ali Mohammad Nejad Sigaroudi, Quantification of Transition Metals in Patients at the Cologne University Hospital, University of Cologne
Other Study IDs: KPUK-14-Metal
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Neurodegenerative Diseases; Infections
MeSH Terms: conditions — Neurodegenerative Diseases; Infections

STUDY DESIGN:
Observational Model: Ecologic or Community
Biospecimen Retention: Samples Without DNA — Remaining portions of samples collected for diagnostic or therapeutic reasons (paired CSF and blood serum samples). No lumbar puncture will be done specifically for this protocol.

GROUPS / COHORTS (4):
- Patients with Parkinson´s Disease
- Patient´s with Alzheimer´s Disease
- Patients with Multiple Sclerosis
- Patients with any other neurodegenerative diseases

SUMMARY:
In this trial, concentrations of transition metals of interest are quantified in surplus cerebrospinal fluid (CSF) and blood serum samples. Quantification of the transition metals will be performed by inductively coupled plasma mass spectrometry (ICP-MS). The treating physicians as well as the patients will not be informed about the results of drug concentrations.

DETAILED DESCRIPTION:
Samples used include:

Remaining portions of samples collected for diagnostic or therapeutic reasons (paired CSF and blood serum samples). No lumbar puncture will be done specifically for this protocol.

The objective of this study is to gain an overview about transition metals concentrations in blood serum and CSF in order to provide preliminary data on patients. The effect of neurodegenerative diseases on metals or the other way round will be assessed if possible.

ELIGIBILITY:
Inclusion Criteria: •

* The trial will include any patient (with various diseases, especially neurodegenerative diseases) who received a lumbar puncture.

Exclusion Criteria:

* • The lower age limit is 18 years. In concordance with the objective of the project there is no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: neurodegenerative diseases infections
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Transition metal concentration | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacology, Cologne, North Rhine-Westphalia, Germany